CLINICAL TRIAL: NCT04695301
Title: Functional Outcomes in COVID-19 Survivors and Use of a Digital Platform for Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 34170820.0.1001.0071
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Coronavirus Infections; Exercise Therapy
Keywords: Telemedicine; exercise therapy; coronavirus infections; stress disorders traumatic; fatigue; quality of life
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Stress Disorders, Traumatic; Fatigue

STUDY DESIGN:
Intervention Model Description: Men and women affected by COVID-19, over 18 years of age, admitted to HIAE partner hospitals who have been in hospital for more than 10 days or in need of treatment in semi-intensive or intensive care units will be selected. Follow-up will be carried out for 3 months, with remote reevaluations. During this period, the rehabilitation program will be offered for 3 months, through a digital platform.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital platform rehabilitation (Experimental): Rehabilitation program through a digital platform for 3 months
  Interventions: Other: Rehabilitation protocol through a digital platform
- control group (Experimental): Patients without access to technology will do the exercises using booklets and will compose the control group
  Interventions: Other: Rehabilitation protocol through a digital platform

INTERVENTIONS:
Other: Rehabilitation protocol through a digital platform — During 3 months the patients will participate in a rehabilitation program through a digital platform

SUMMARY:
COVID-19, an acute respiratory disease caused by coronavirus-2 (SARS-CoV-2), and in most cases, causes mild to moderate symptoms of fever, cough and dyspnea. However, a not insignificant portion, given the total number of people affected, will present symptoms of severe acute respiratory failure and multiple organ failure, requiring hospitalization under intensive care, use of mechanical ventilation, prolonged period of immobilization and, consequently, physical, cognitive and psychological damage, which may affect survivors for a long period after hospitalization. All of these factors are known to have an impact on various areas of life: personal, social and economic, which makes the need for continued specific care after hospital discharge relevant. In this context, the role of rehabilitation programs is fundamental, aiming not only at a safer dehospitalization, but also at the continuity of care with the objective of restoring the biopsychosocial skills of these individuals, allowing functional independence for activities of daily life and a shorter return physical and social activities performed before the disease. However, the big challenge for the health system is how to offer this on a large scale. Therefore, knowing the clinical and functional profile of these patients at discharge and verifying the viability of a digital platform for rehabilitation and monitoring of these patients is the first step to allow the creation of a new form of continuity of care and access to affected patients with serious diseases such as COVID-19 and other syndromes capable of generate functional impairment. Therefore,the investigators objective is to characterize and monitor the functional profile and exercise capacity of patients affected by COVID-19 at the hospital discharge, as well as to verify the viability and compliance of patients to the use of a digital platform for the application of a distance rehabilitation program.

DETAILED DESCRIPTION:
The investigators proposal is to characterize and evaluate the impact of the disease on the clinical, functional and social aspects in these patients affected by COVID-19 and to propose the continuity of specific care after hospital discharge with a physical rehabilitation program through a digital platform, remotely for a period of 3 months. The proposed hypothesis is that patients convalescing from COVID-19 and undergoing the rehabilitation program will have a gain in functional skills and quality of life. The professional team involved in this study will be responsible for managing, monitoring and evaluating the participating patients and monitoring the performance of the proposed functional exercises.

ELIGIBILITY:
Inclusion Criteria:

* Men and women affected by COVID-19
* over 18 years of age, admitted to HIAE partner hospitals

Exclusion Criteria:

* presence of a physical or cognitive condition that makes it impossible or contraindicated to perform the 2-minute stride test and perform the proposed exercises.
* Patients with a more severe clinical and functional profile,
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Characterize the clinical function profile of patients affected by COVID-19 | 3 months
  Characterize the clinical functional profile of patients affected by COVID-19 by data from medical records
Characterize the exercise capacity of patients affected by COVID-19 | 3 months
  Characterize the exercise capacity of patients affected by COVID-19 by 2-minute step test

SECONDARY OUTCOMES:
Assess clinical and demographic data | 3 months
  Assess clinical and demographic data
Assess functional level at hospital discharge | 3 months
  Assess functional level at hospital discharge and 3 months after discharge by physical test
Assess patient compliance of the rehabilitation program using the digital platform | 3 months
  Assess patient compliance of the rehabilitation program using the digital platform checking your adherence to the program

CONTACTS AND LOCATIONS:
Overall Officials: Luciana D Matos, MD,PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein 's (IIEP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: when to published